CLINICAL TRIAL: NCT00561691
Title: Phase III Study on the Effectiveness of OSAG 101 (Theraloc®)in Newly Diagnosed Intrinsic Pontine Gliomas of Children and Adolescents
Brief Title: Nimotuzumab in Children With Intrinsic Pontine Glioma
Status: Completed | Type: Observational
Sponsor: Oncoscience AG (Industry)
Collaborators: Children's Medical Hospital, University of Bonn, Germany (Other); University of Wuerzburg (Other); Dept. of Statistics, University of Dortmund, Germany (Other); CRM Biometrics GmbH (Industry); Heinrich-Heine University, Duesseldorf (Other); Dr. von Haunersches Children's Medical Hospital, University of Munich, Germany (Other); Children's Medical Hospital, University of Homburg/Saar, Homburg/Saar, Germany (Other); Children's Medical Hospital, Medical School Hannover, Hannover, Germany (Unknown); Children's Medical Hospital, University of Leipzig, Leipzig, Germany (Other); Children's Medical Hospital, University of Muenster, Muenster, Germany (Other); Burdenko Neurosurgery Institute (Other); Istituto Nazinonale Tumori, Div. of Paediatric Oncology,Milano, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: OSAG101-BSC05
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Diffuse Instrinsic Ponitine Glioma
Keywords: diffuse instrinsic ponitine glioma, brainstem
MeSH Terms: interventions — nimotuzumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: nimotuzumab — monoclonal antibody
  Other Names: Theraloc

SUMMARY:
Determination of efficiency of nimotuzumab in children with diffuse intrinsic pontine glioma.

DETAILED DESCRIPTION:
Due to the poor prognosis of diffuse intrinsic pontine gliomas, the limited therapy options, the relevant portion of EGFR expression and the unexpected good response to the therapy with OSAG 101 in the phase II study, a phase III study was planned in newly diagnosed diffuse intrinsic pontine gliomas in children and adolescents. A phase II study in patients of recurrence/resistance high grade glioma in childhood or adolescence showed that, in particular, a part of the intrinsic pontine glioma response to the monotherapy with OSAG 101 resulting in a reduction in the size of the tumour or stabilisation in the growth of the tumour. Together with clinical improvement, stabilisation lasted markedly over 6 months in two thirds of the patients. The current phase III study was scheduled to provide evidence of the effectiveness in the case of newly diagnosed intrinsic pontine glioma. In this study, OSAG 101 will be given concomitantly to the only standard therapy for this kind of tumour, i.e. the fractionated radiotherapy, to show effectiveness in the primary endpoint of median progression-free survival, the secondary endpoint of median overall survival and the side effect profile.

Evidence from the median progression-free survival and the side effect profile of this combination met the expected results and one may consider that combination therapy of this therapeutic approach with other immunotherapeutic or antiangiogenic approaches and/or mild chemotherapy could lead to a better prognosis and quality of life for these patients.

ELIGIBILITY:
Inclusion Criteria:

Histology and staging of disease:

* Newly diagnosed intrinsic pontine glioma documented by MRI and measurable in at least one dimension
* Histology is not required for this study, tumour biopsy is not recommended General conditions
* Age ≥ 3 years to ≤ 20 years, both gender
* Life expectancy ≥ 4 weeks
* Performance status ECOG ≥ 3 or Karnofsky/Lansky status ≥ 40%
* Adequate haematological, renal, and hepatic function Absolute leukocyte count ≥ 2.0 x 109/l Haemoglobin ≥ 10 g/dl Platelets ≥ 50 x 109/l Bilirubin total ≤ 2.5 x ULN ALT/AST ≤ 5.0 x ULN Creatinine i. S. ≤ 1.5 x ULN

Prior/initial examinations (within 14 days prior to the start of therapy):

* Cranial MRI (estimation of index lesion)
* Clinical internal and neurological examination; body weight, height, surface, Performance status by ECOG, Karnofsky or Lansky
* Blood cell count, blood gas analysis; serum analysis for electrolytes (Na, K, Ca, Mg), chloride, phosphate, creatinine, BUN, AST, ALT, bilirubin, GGT, LDH, lipase, total protein, CRP, blood sugar; coagulation test (Quick, PTT, TT); urinalysis
* EKG, echocardiography in case of positive cardiac history
* Pregnancy test in females of childbearing age Other criteria
* Planned day of first antibody application within 14 days after MRI
* Written and signed informed consent from patient and/or parents or legal guardian(s)(s) after being informed
* Negative pregnancy test in females of childbearing age
* Treatment in a study centre
* Availability of the patient during the study treatment and the ability to comply with the study plan

Exclusion Criteria:

* Pontine glioma as secondary malignancy
* Low grade brain stem glioma (i.e. focal, cervicomedullar, tectal brain stem glioma)
* Other severe underlying disease or pre-existing serious conditions which bear the risk of an inadequate study treatment (e.g. severe mental retardation, severe statomotoric retardation, severe cerebral palsy, congenital syndromes)
* Prior antineoplastic therapy, inclusively chemotherapy, immunotherapy, radiotherapy
* Prior administration of a recombinant human or mural antibody or known hypersensitivity to antibodies
* Simultaneous antineoplastic therapy other than the study treatment
* Participation in another therapeutic study or experimental treatment involving the underlying cancer disease
* Pregnancy, lactating mother and inadequate contraception in females and males of childbearing age

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children and adolescents
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2006-04; Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To determine the progression-free survival (PFS) of the combination of monoclonal anti-EGFR antibody OSAG 101 and standard local radiotherapy | week 12, 24, 36

SECONDARY OUTCOMES:
To determine the objective response rate (R=CR+PR+SD/Nr) according to RECIST To determine the duration of response and the overall survival To assess adverse events and the toxicity profile according to CTCAE version 3.0 | week 12, 24, 36

CONTACTS AND LOCATIONS:
Overall Officials: Udo Bode, Prof. MD, Principal Investigator — University Bonn
Locations (1):
- University Bonn, Children's Medical Hospital, Bonn, Germany

REFERENCES:
- See also: Related Info — http://ukb.uni-bonn.de